CLINICAL TRIAL: NCT02063412
Title: The Impact of Nursing and Pharmacy Care Between Capecitabine and 5-Fluoruracil Regimens in the Management of Advanced Esophago-gastric Cancer in Hong Kong
Brief Title: Nursing and Pharmacy Care Between Capecitabine and 5-Fluoruracil Regimens
Status: Withdrawn | Type: Observational
Why Stopped: Slow recruitment pace
Sponsor: Vivian Wing Yan Lee (Other)
Collaborators: Hoffmann-La Roche (Industry); Queen Elizabeth Hospital, Hong Kong (Other); Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Sponsor-Investigator, Vivian Wing Yan Lee, Associate Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: Roche-TR116583; TR116583VLKZ003 (Other: CUHK)
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- XELOX: Capecitabine (Xeloda) 1000mg/m2 po bid x 14 days Oxaliplatin (Eloxatin) 130mg/m2 iv over 2 hrs d1 Q3w x 8 cycles
- XP: Cisplatin (CDDP) 80 mg/m2 iv over 3 hrs d1 Capecitabine (Xeloda) 1000 mg/m2 po bid d1-14, Q3w
- FOLFOX: Leucovorin 200 mg/m2 iv over 2 hrs before 5-FU, d1 and d2 5-FU 400mg/m2 iv bolus and then 600 mg/m2 iv over 22 hrs, d1 and d2 Q2w
- FP: Cisplatin (CDDP) 100 mg/m2 iv d1 5-FU 1000 mg/m2/d civi d1-5, Q4w

SUMMARY:
The objective of this study is to compare the possible time savings from reduction of nursing and pharmacy time to manage AEGC patients using capecitabine-based regimens versus traditional intravenous chemotherapy in the Hong Kong public hospital setting.

DETAILED DESCRIPTION:
Advanced esophageal and gastric cancer (AEGC) have ranked in the top 10 cancer-related cause of death worldwide, with approximately one million new cases each year. Over half of new cases are in East Asia. The traditional chemotherapy for AEGC remains on intravenous (IV) fluorouracil (5-FU), cisplatin, and the anthracyclines. Trials favoured the combined use of 5-FU and cisplatin for superior efficacy and quality of life in AEGC patients. Recent years, oral chemotherapy has a more practical and economic advantages over IV regimen. It is understandable that patients prefer oral regimens as long as the clinical efficacy is maintained. Oral treatment strategy preserves quality of life for AEGC patients. In addition, it may also have additional cost saving in the nursing and pharmacy time. It is because a significant amount of time can be saved in both nursing and pharmacy for the preparation and administration of IV chemotherapy However, there is a lack of local data to demonstrate the impact of pharmacy and nursing care utilizing capecitabine-based regimen comparing to traditional IV chemotherapy in MCRC patients of Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above
2. Diagnosed with AEGC and were prescribed with either XELOX-based or FOLFOX4- based chemotherapy treatment

Exclusion Criteria:

1. Persons < 18 years of age;
2. Pregnant or lactating women;
3. Persons related unequally to investigators (e.g. student, employee);
4. Special population (e.g. prisoner, mentally, congnitively disabled);
5. Patients who refused to sign consent or not willing to participate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were diagnosed with AEGC and were prescribed with either XELOX-based or FOLFOX4-based chemotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Composite preparation, dispensing, and administration time | Up to 6 months after initiation of chemotherapy
  This is a time-and-motion study conducted in 2 public hospitals of Hong Kong based on the simulation of previously data on both capecitabine-based regimen (XELOX and XP) and IV 5-FU-based regimen (FOLFOX and FP)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian WY Lee, PharmD, Principal Investigator — Chinese University of Hong Kong